CLINICAL TRIAL: NCT02485691
Title: A Randomized, Open Label, Multicenter Study of Cabazitaxel Versus an Androgen Receptor (AR)-Targeted Agent (Abiraterone or Enzalutamide) in mCRPC Patients Previously Treated With Docetaxel and Who Rapidly Failed a Prior AR-targeted Agent (CARD)
Brief Title: Cabazitaxel Versus the Switch to Alternative AR-targeted Agent (Enzalutamide or Abiraterone) in Metastatic Castration-resistant Prostate Cancer (mCRPC) Patients Previously Treated With Docetaxel and Who Rapidly Failed a Prior AR-targeted Agent
Acronym: CARD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPS14201; 2014-004676-29 (EudraCT Number); U1111-1166-5329 (Other: UTN)
Record Dates: First submitted 2015-06-26; First posted 2015-06-30 (Estimated); Results first posted 2022-02-14 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Prostate Cancer Metastatic
MeSH Terms: interventions — cabazitaxel; enzalutamide; Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cabazitaxel (Experimental): Participants received Cabazitaxel 25 mg/m^2 intravenous (IV) infusion for over 1 hour on Day 1 of each 3 week treatment cycle in combination with Prednisone 10 mg orally once daily and primary prophylactic granulocyte-colony stimulating factor (G-CSF) as per investigator decision, until radiographic disease progression, unacceptable toxicity, or participant's refusal of further study treatment (median duration = 22 weeks).
  Interventions: Drug: cabazitaxel XRP6258; Drug: prednisone
- Abiraterone acetate or enzalutamide (Experimental): Participants received either abiraterone acetate 1000 mg orally once daily from Day 1 to Day 21 of each 3 week treatment cycle in combination with prednisone 5 mg orally twice daily; or enzalutamide 160 mg orally once daily continuously from Day 1 to Day 21 of each 3 week treatment cycle, until radiographic disease progression, unacceptable toxicity, or participant's refusal of further study treatment (median duration = 12.5 weeks).
  Interventions: Drug: enzalutamide; Drug: abiraterone acetate; Drug: prednisone

INTERVENTIONS:
Drug: cabazitaxel XRP6258 — Pharmaceutical form: solution Route of administration: intravenous
  Other Names: Jevtana
  Arms: Cabazitaxel
Drug: enzalutamide — Pharmaceutical form: capsule Route of administration: oral
  Other Names: Xtandi
  Arms: Abiraterone acetate or enzalutamide
Drug: abiraterone acetate — Pharmaceutical form: tablet Route of administration: oral
  Other Names: Zytiga
  Arms: Abiraterone acetate or enzalutamide
Drug: prednisone — Pharmaceutical form: tablet Route of administration: oral

SUMMARY:
Primary Objective:

To compare the radiographic progression-free survival (rPFS) (using Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 for tumor lesions and Prostate Cancer Working Group 2 (PCWG2) criteria for bone scan lesions or death due to any cause) with chemotherapy (cabazitaxel plus prednisone, Arm A) versus Androgen Receptor (AR)-targeted therapy (enzalutamide or abiraterone acetate plus prednisone, Arm B) in mCRPC participants who have been treated with docetaxel and who had disease progression while receiving AR-targeted therapy within 12 months of AR treatment initiation (less than or equal to [<=]12 months, either before or after docetaxel).

Secondary Objective:

* To compare efficacy for:
* Prostate-specific antigen (PSA) response rate and time to PSA progression (TTPP).
* Progression-free survival (PFS).
* Overall survival (OS).
* Tumor response rate and duration of tumor response.
* Pain response and time to pain progression.
* Symptomatic skeletal event (SSE) rate and time to occurrence of any SSE.
* Health status and Health-related Quality of Life (HRQOL).
* To evaluate the correlation of a signature of resistance to AR-targeted agents with clinical outcome via the analysis of circulating tumor cell (CTC) phenotypes as well as expression and localization of proteins including AR isoforms in CTCs.
* To evaluate safety in the 2 treatment arms.

DETAILED DESCRIPTION:
The duration of the study per participant was approximately 2 years. Each participant was treated until radiographic disease progression, unacceptable toxicity, or participant's refusal of further study treatment, and each participant was followed after completion of study treatment until death, study cut-off date, or withdrawal of participant consent.

ELIGIBILITY:
Inclusion criteria :

Histologically confirmed prostate adenocarcinoma.

* Metastatic disease.
* Effective castration with serum testosterone levels less than (<)0.5 ng/mL. If the participant has been treated with Luteinizing hormone-releasing hormone agonist (LHRH) agonists or antagonist (i.e., without orchiectomy), then this therapy should be continued.
* Progressive disease defined by at least one of the following:
* Progression in measurable disease (RECIST 1.1 criteria).
* Appearance of 2 or more new bone lesions (PCWG2).
* Rising Prostate Specific Antigen (PSA) (PCWG2).
* Having received prior docetaxel for at least 3 cycles (before or after an AR-targeted therapy). Docetaxel administration in combination with androgen deprivation therapy (ADT) in metastatic hormone-sensitive disease was considered a prior exposure. Docetaxel rechallenge was allowed.
* Having progressive disease (PD) while receiving AR-targeted therapy with abiraterone acetate or enzalutamide within 12 months of AR treatment initiation (<=12 months), even if treatment duration was longer than 12 months. Participants treated with Abiraterone Acetate + ADT in metastatic hormone-sensitive setting were eligible in the study if they have progressed within 12 months with the AR-targeted agent. Participants having PSA progression only (as per PCWG2) within 12 months were eligible.
* A PSA value of at least 2 ng/mL was required at study entry.
* Prior AR-targeted therapy (abiraterone acetate or enzalutamide) must be stopped at least 2 weeks before study treatment.
* Signed informed consent.

Exclusion criteria:

* Prior chemotherapy other than docetaxel for prostate cancer, except estramustine and except adjuvant/neoadjuvant treatment completed >3 years ago.
* Less than 28 days elapsed from prior treatment with chemotherapy, immunotherapy, radiotherapy, or surgery to the time of randomization.
* Adverse events (excluding alopecia and those listed in the specific exclusion criteria) from any prior anticancer therapy of Grade >1 (National Cancer Institute Common Terminology Criteria [NCI CTCAE] v4.0) at the time of randomization.
* Eastern Cooperative Oncology Group performance status (ECOG PS) >2 (ECOG 2 must be related to prostate cancer, not to other comorbidities).
* Prior malignancy. Adequately treated basal cell or squamous cell skin or superficial (pTis, pTa, and pT1) bladder cancer were allowed, as well as any other cancer for which treatment has been completed >=5 years ago and from which the participant has been disease-free for >=5 years.
* Participation in another clinical trial and any concurrent treatment with any investigational drug within 30 days prior to randomization.
* Acquired immunodeficiency syndrome (AIDS-related illnesses) or known human immunodeficiency virus (HIV) disease requiring antiretroviral treatment.
* Participants with reproductive potential who do not agree, in conjunction with their partner, to use accepted and effective method of contraception during the study treatment period and up to 6 months after the last administered dose. The definition of "effective method of contraception" described hereafter: oral contraceptives, combined hormonal intravaginal, transdermal, intra uterine device or condoms was based on respective study treatment labelling and country-specific regulatory requirements, and were documented in the Informed Consent Form.
* Known allergies, hypersensitivity or intolerance to prednisone or excipients of abiraterone acetate, enzalutamide, docetaxel, or polysorbate 80.
* Known history of mineralocorticoid excess or deficiency.
* History of seizure, underlying brain injury with loss of consciousness, transient ischemic attack within the past 12 months, cerebral vascular accident, brain arteriovenous malformation, brain metastases, or the use of concomitant medications that may lower the seizure threshold.
* Unable to swallow a whole tablet or capsule.
* Inadequate organ and bone marrow function as evidenced by:
* Hemoglobin <10.0 g/dL;
* Absolute neutrophil count <1.5 * 10^9/L;
* Platelet count <100 * 10^9/L;
* Aspartate aminotransferase/serum glutamic oxaloacetic transaminase and/or alanine aminotransferase/serum glutamic pyruvic transaminase >1.5 * the upper limit of normal (ULN);
* Total bilirubin >1.0 * ULN;
* Potassium <3.5 mmol/L;
* Child-Pugh Class C.
* Contraindications to the use of corticosteroid treatment.
* Symptomatic peripheral neuropathy Grade >=2 (NCI CTCAE v4.0).
* Uncontrolled severe illness or medical condition including uncontrolled diabetes mellitus, history of cardiovascular disease (uncontrolled hypertension, arterial thrombotic events in the past 6 months, congestive heart failure, severe or unstable angina pectoris, recent myocardial infarction within the last 6 months, or uncontrolled cardiac arrhythmia).
* Concomitant vaccination with yellow fever vaccine.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2015-11-09 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2021-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (65):
- Austria (3):
  - Investigational Site Number 040002, Linz
  - Investigational Site Number 040003, Vienna
  - Investigational Site Number 040004, Vienna
- Belgium (6):
  - Investigational Site Number 056013, Bruges
  - Investigational Site Number 056003, Brussels
  - Investigational Site Number 056007, Brussels
  - Investigational Site Number 056006, Charleroi
  - Investigational Site Number 056001, Ghent
  - Investigational Site Number 056005, Leuven
- Czechia (4):
  - Investigational Site Number 203005, Brno
  - Investigational Site Number 203001, Olomouc
  - Investigational Site Number 203002, Pilsen
  - Investigational Site Number 203003, Prague
- France (14):
  - Investigational Site Number 250010, Clermont-Ferrand
  - Investigational Site Number 250006, Lyon
  - Investigational Site Number 250004, Marseille
  - Investigational Site Number 250011, Montpellier
  - Investigational Site Number 250013, Paris
  - Investigational Site Number 250007, Paris
  - Investigational Site Number 250002, Paris
  - Investigational Site Number 250014, Plérin
  - Investigational Site Number 250016, Reims
  - Investigational Site Number 250018, Saint-Mandé
  - Investigational Site Number 250009, Strasbourg
  - Investigational Site Number 250005, Suresnes
  - Investigational Site Number 250008, Tours
  - Investigational Site Number 250001, Villejuif
- Germany (14):
  - Investigational Site Number 276028, Aschaffenburg
  - Investigational Site Number 276008, Berlin
  - Investigational Site Number 276022, Duisburg
  - Investigational Site Number 276023, Essen
  - Investigational Site Number 276002, Frankfurt am Main
  - Investigational Site Number 276007, Göttingen
  - Investigational Site Number 276026, Jena
  - Investigational Site Number 276025, Lübeck
  - Investigational Site Number 276004, Magdeburg
  - Investigational Site Number 276018, Mannheim
  - Investigational Site Number 276006, Münster
  - Investigational Site Number 276003, Nürtingen
  - Investigational Site Number 276010, Rostock
  - Investigational Site Number 276011, Tübingen
- Greece (3):
  - Investigational Site Number 300001, Athens
  - Investigational Site Number 300005, Marousi, Athens
  - Investigational Site Number 300004, Thessaloniki
- Investigational Site Number 352001, Reykjavik, Iceland
- Ireland (2):
  - Investigational Site Number 372001, Dublin
  - Investigational Site Number 372003, Dublin
- Italy (7):
  - Investigational Site Number 380004, Brescia
  - Investigational Site Number 380005, Candiolo
  - Investigational Site Number 380009, Meldola
  - Investigational Site Number 380006, Napoli
  - Investigational Site Number 380002, Pisa
  - Investigational Site Number 380001, Roma
  - Investigational Site Number 380008, Verona
- Netherlands (4):
  - Investigational Site Number 528002, Breda
  - Investigational Site Number 528003, Nijmegen
  - Investigational Site Number 528005, Rotterdam
  - Investigational Site Number 528004, Sittard-Geleen
- Norway (2):
  - Investigational Site Number 578001, Grålum
  - Investigational Site Number 578002, Trondheim
- Spain (4):
  - Investigational Site Number 724001, Barcelona
  - Investigational Site Number 724004, Madrid
  - Investigational Site Number 724002, Madrid
  - Investigational Site Number 724003, Seville
- Investigational Site Number 826001, Sutton, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Longoria O, Rekowski J, Gupta S, Beije N, Pantel K, Efstathiou E, Sternberg C, Castellano D, Fizazi K, Tombal B, Sharp A, Sartor O, Mace S, Geffriaud-Ricouard C, Wenstrup R, de Wit R, de Bono J. Chromosomal instability in circulating tumor cells and cabazitaxel resistance in metastatic castration-resistant prostate cancer. JCI Insight. 2025 Nov 4;10(24):e196505. doi: 10.1172/jci.insight.196505. eCollection 2025 Dec 22. PMID 41186991
- [Derived] de Wit R, Wulfing C, Castellano D, Kramer G, Eymard JC, Sternberg CN, Fizazi K, Tombal B, Bamias A, Carles J, Iacovelli R, Melichar B, Sverrisdottir A, Theodore C, Feyerabend S, Helissey C, Foster MC, Ozatilgan A, Geffriaud-Ricouard C, de Bono J. Baseline neutrophil-to-lymphocyte ratio as a predictive and prognostic biomarker in patients with metastatic castration-resistant prostate cancer treated with cabazitaxel versus abiraterone or enzalutamide in the CARD study. ESMO Open. 2021 Oct;6(5):100241. doi: 10.1016/j.esmoop.2021.100241. Epub 2021 Aug 24. PMID 34450475
- [Derived] Sternberg CN, Castellano D, de Bono J, Fizazi K, Tombal B, Wulfing C, Kramer G, Eymard JC, Bamias A, Carles J, Iacovelli R, Melichar B, Sverrisdottir A, Theodore C, Feyerabend S, Helissey C, Poole EM, Ozatilgan A, Geffriaud-Ricouard C, de Wit R. Efficacy and Safety of Cabazitaxel Versus Abiraterone or Enzalutamide in Older Patients with Metastatic Castration-resistant Prostate Cancer in the CARD Study. Eur Urol. 2021 Oct;80(4):497-506. doi: 10.1016/j.eururo.2021.06.021. Epub 2021 Jul 15. PMID 34274136
- [Derived] Fizazi K, Kramer G, Eymard JC, Sternberg CN, de Bono J, Castellano D, Tombal B, Wulfing C, Liontos M, Carles J, Iacovelli R, Melichar B, Sverrisdottir A, Theodore C, Feyerabend S, Helissey C, Oudard S, Facchini G, Poole EM, Ozatilgan A, Geffriaud-Ricouard C, Bensfia S, de Wit R. Quality of life in patients with metastatic prostate cancer following treatment with cabazitaxel versus abiraterone or enzalutamide (CARD): an analysis of a randomised, multicentre, open-label, phase 4 study. Lancet Oncol. 2020 Nov;21(11):1513-1525. doi: 10.1016/S1470-2045(20)30449-6. Epub 2020 Sep 11. PMID 32926841
- [Derived] de Wit R, de Bono J, Sternberg CN, Fizazi K, Tombal B, Wulfing C, Kramer G, Eymard JC, Bamias A, Carles J, Iacovelli R, Melichar B, Sverrisdottir A, Theodore C, Feyerabend S, Helissey C, Ozatilgan A, Geffriaud-Ricouard C, Castellano D; CARD Investigators. Cabazitaxel versus Abiraterone or Enzalutamide in Metastatic Prostate Cancer. N Engl J Med. 2019 Dec 26;381(26):2506-2518. doi: 10.1056/NEJMoa1911206. Epub 2019 Sep 30. PMID 31566937

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 66 active centers in 13 countries. A total of 255 participants were randomized between 09 November 2015 to 13 November 2018, out of which 250 participants received treatment with the study drug.
Pre-assignment Details: Participants were randomized to receive either cabazitaxel or Androgen receptor (AR) targeted therapy (abiraterone or enzalutamide were assigned based on previous AR targeted treatment in which participants previously treated with abiraterone were treated with enzalutamide and vice versa due to resistance).
Groups:
- Abiraterone Acetate or Enzalutamide: Participants received either abiraterone acetate 1000 mg orally once daily from Day 1 to Day 21 of each 3 week treatment cycle in combination with prednisone 5 mg orally twice daily; or enzalutamide 160 mg orally once daily continuously from Day 1 to Day 21 of each 3 week treatment cycle, until radiographic disease progression, unacceptable toxicity, or participant's refusal of further study treatment (median duration =12.5 weeks)
Period: Overall Study
Arm/Group | Cabazitaxel | Abiraterone Acetate or Enzalutamide
Started | 129 | 126
Treated | 126 | 124
Completed | 0 | 0
Not Completed | 129 | 126
Not completed — Adverse Event | 25 | 11
Not completed — Poor compliance to protocol | 0 | 1
Not completed — Disease progression | 57 | 92
Not completed — Investigator's decision | 23 | 5
Not completed — Participant's request | 13 | 6
Not completed — Other reason | 8 | 9
Not completed — Randomized and not treated | 3 | 2

BASELINE CHARACTERISTICS:
Population: Analysis was performed on Intent-to-treat (ITT) population, that included any participant who had been allocated to a randomized treatment regardless of whether the treatment kit was used, analyzed according to the treatment group allocated by randomization.
Groups:
- Cabazitaxel: Participants received Cabazitaxel 25 mg/m^2 IV infusion for over 1 hour on Day 1 of each 3 week treatment cycle in combination with Prednisone 10 mg orally once daily and primary prophylactic G-CSF as per investigator decision, until radiographic disease progression, unacceptable toxicity, or participant's refusal of further study treatment (median duration = 22 weeks).
- Total: Total of all reporting groups
Arm/Group | Cabazitaxel | Abiraterone Acetate or Enzalutamide | Total
Number analyzed (Participants) | 129 | 126 | 255
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (8.3) | 69.7 (7.9) | 69.7 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 129 | 126 | 255
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Progression-Free Survival (rPFS)
Description: Radiographic progression-free survival: time (in months) from randomization to occurrence of any one of following: radiological tumor progressions using response evaluation criteria in solid tumors (RECIST 1.1), progression of bone lesions using Prostate Cancer Working Group 2 (PCWG2) criteria or occurrence of death due to any cause. Progression as per RECIST 1.1: at least a 20 percent (%) increase in sum of diameters of target lesions, unequivocal progression of existing non-target lesions. Progression of bone lesions (PCWG2 criteria): first bone scan with >= 2 new lesions compared to Baseline observed less than (<) 12 weeks from randomization and confirmed by a second bone scan performed >=6 weeks; first bone scan with >=2 new lesions compared to Baseline observed >=12 weeks from randomization. In accordance with protocol, data cut-off date for final analysis of this endpoint was the date when 196 rPFS events had occurred. Analysis done by Kaplan-Meier method.
Time Frame: From randomization until tumor progression or bone lesion progression, death due to any cause, or data cut-off date whichever comes first (maximum duration: up to 141 weeks)
Population: Analysis was performed on ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabazitaxel | Abiraterone Acetate or Enzalutamide
Number analyzed (Participants) | 129 | 126
months | 8.0 [5.7 to 9.2] | 3.7 [2.8 to 5.1]
Statistical Analysis 1: Comparison: Cabazitaxel vs Abiraterone Acetate or Enzalutamide; Hazard ratio was estimated using a Cox Proportional Hazards regression model. The Cox proportional hazard model was stratified by ECOG performance status, time from AR- targeted agent initiation progression, timing of AR targeted agent as specified at the time of randomization; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error. Testing was then performed sequentially in order the outcome measure are reported and continued when previous outcome measure was statistically significant at two-sided 0.05. Only the primary and the first 4 secondary outcome measures were included in the procedure; p < 0.0001, Log Rank — P-value from 2-sided stratified log-rank test, stratified for ECOG performance status, time from AR- targeted agent initiation progression, timing of AR targeted agent as specified at the time of randomization. Significance threshold was at 0.05; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.40 to 0.73] — Cabazitaxel vs Abiraterone Acetate or Enzalutamide

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time interval (in months) from the date of randomization to the date of death due to any cause. In the absence of confirmation of death, survival time was censored at the last date participant was known to be alive, or at the cut-off date whichever comes first. Analysis was performed by Kaplan-Meier method.
Time Frame: From randomization to death due to any cause, or data cut-off date whichever comes first (maximum duration: up to 141 weeks)
Population: Analysis was performed on ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabazitaxel | Abiraterone Acetate or Enzalutamide
Number analyzed (Participants) | 129 | 126
months | 13.6 [11.5 to 17.5] | 11.0 [9.2 to 12.9]
Statistical Analysis 1: Comparison: Cabazitaxel vs Abiraterone Acetate or Enzalutamide; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0078, Log Rank — P-value from two-sided stratified log-rank test, stratified for ECOG performance status, time from AR-targeted agent initiation to progression, timing of AR-targeted agent as specified at the time of randomization. Significance threshold = 0.05; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.46 to 0.89] — Cabazitaxel vs Abiraterone Acetate or Enzalutamide

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS:time duration (in months) from date of randomization to date of first occurrence of any of following events: radiological tumor progression (RECIST 1.1); progression of bone lesions (PCWG2); symptomatic progression (developing urinary or bowel symptoms; need to change anti-cancer therapy), pain progression or death due to any cause. Tumor Progression(RECIST 1.1): at least 20% increase in sum of diameters of target lesions, unequivocal progression of existing non-target lesions. Progression of bone lesion (PCWG2 criteria): first bone scan with >=2 new lesions compared to Baseline and confirmed by second bone scan performed >=6 weeks later; pain progression: increase by >=30% from Baseline in pain intensity score (calculated using scale ranged from 0=no pain to 5=extreme pain) or increase in analgesic usage score >=30% (calculated from analgesic use data, non-narcotic medications assigned value of 1 point and narcotic medications assigned 4 points). Analyzed by Kaplan-Meier method.
Time Frame: From randomization until tumor progression or bone lesion progression, pain progression, death due to any cause, or data cut-off date whichever comes first (maximum duration: up to 141 weeks)
Population: Analysis was performed on ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabazitaxel | Abiraterone Acetate or Enzalutamide
Number analyzed (Participants) | 129 | 126
months | 4.4 [3.6 to 5.4] | 2.7 [2.3 to 2.8]
Statistical Analysis 1: Comparison: Cabazitaxel vs Abiraterone Acetate or Enzalutamide; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.40 to 0.68] — Cabazitaxel vs Abiraterone Acetate or Enzalutamide

4. Secondary Outcome: Percentage of Participants With Prostate Specific Antigen (PSA) Response
Description: PSA response was defined as >= 50% decrease from baseline in serum PSA levels, confirmed by a second PSA value at least 3 weeks later.
Time Frame: Baseline up to PSA response, death due to any cause or data cut-off date whichever comes first (maximum duration: up to 141 weeks)
Population: Analysis was performed on subset of ITT population (any participant who had been allocated to a randomized treatment, analyzed according to group allocated) with PSA level >2 ng/mL at baseline, and with at least two post-baseline assessments before any further anti-cancer therapy for specified outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cabazitaxel | Abiraterone Acetate or Enzalutamide
Number analyzed (Participants) | 113 | 105
percentage of participants | 36.3 [27.4 to 45.1] | 14.3 [7.6 to 21.0]
Statistical Analysis 1: Comparison: Cabazitaxel vs Abiraterone Acetate or Enzalutamide; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0003, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel test stratified by ECOG performance status, time from AR-targeted agent initiation to progression, timing of AR-targeted agent as specified at the time of randomization. Significance threshold = 0.05

5. Secondary Outcome: Percentage of Participants With Overall Objective Tumor Response
Description: Overall objective tumor response was defined as having a partial response (PR) or complete response (CR) according to the RECIST version 1.1. CR was defined as disappearance of all target and non-target lesions and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From randomization until disease progression, death due to any cause or data cut-off date whichever comes first (maximum duration: up to 141 weeks)
Population: Analysis was performed on subset of ITT population (any participant who had been allocated to a randomized treatment, analyzed according to group allocated) with measurable disease at baseline and at least one post-baseline assessment before any further anti-cancer therapy for specified outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cabazitaxel | Abiraterone Acetate or Enzalutamide
Number analyzed (Participants) | 63 | 52
percentage of participants | 36.5 [24.6 to 48.4] | 11.5 [2.9 to 20.2]
Statistical Analysis 1: Comparison: Cabazitaxel vs Abiraterone Acetate or Enzalutamide; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0004, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]

6. Secondary Outcome: Time to PSA Progression (TTPP)
Description: TTPP was defined as the time duration (in months) between the date of randomization and the date of first documented PSA progression. PSA progression (as per PCWG 2) was defined as: 1) If decline from Baseline value: an increase of >=25% (at least 2 ng/mL) over the nadir value, confirmed by a second PSA value at least 3 weeks apart; 2) If no decline from Baseline value: an increase of >=25% (at least 2 ng/mL) over the baseline value after 12 weeks of treatment, confirmed by a second PSA value at least 3 weeks apart. Analysis performed by Kaplan-Meier method.
Time Frame: From time from randomization until PSA progression, death due to any cause or data cut-off whichever comes first (maximum duration: up to 141 weeks)
Population: Analysis was performed on subset of ITT population (any participant who had been allocated to a randomized treatment, analyzed according to group allocated) with PSA level > 2ng/mL at baseline, and with at least two post-baseline assessments before any further anti-cancer therapy for specified outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabazitaxel | Abiraterone Acetate or Enzalutamide
Number analyzed (Participants) | 113 | 105
months | 6.3 [4.2 to 8.3] | 2.1 [1.7 to 2.3]

7. Secondary Outcome: Duration of Tumor Response
Description: Duration of tumor response was defined as the time (in months) from date of first response (CR or PR) until date of first documentation of tumor progression or death, whichever occurs first. As per RECIST 1.1 CR was defined as disappearance of all target and non-target lesions and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Progression was defined as at least a 20% increase in sum of diameters of target lesions, unequivocal progression of existing non-target lesions. Analysis was performed by Kaplan-Meier method.
Time Frame: From the date of the first response to the date of first documented tumor progression, or death due to any cause or data cut-off date whichever comes first (maximum duration: up to 141 weeks)
Population: Analysis was performed on subset of participants with overall objective tumor response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabazitaxel | Abiraterone Acetate or Enzalutamide
Number analyzed (Participants) | 23 | 6
months | 6.5 [5.6 to 11.4] | 8.0 [1.1 to NA] — Upper limit of Confidence Interval (CI) was not estimable due to less number of participants with overall objective tumor response.

8. Secondary Outcome: Percentage of Participants Achieving Pain Response Assessed Using Brief Pain Inventory-Short Form (BPI-SF) Pain Intensity Score
Description: Pain response as per BPI-SF was defined as a decrease of at least 30% from Baseline in the average of BPI-SF pain intensity score observed at 2 consecutive evaluations >=3 weeks apart without increase in analgesic usage score (calculated from analgesic use data, with non-narcotic medications assigned value of 1 point and narcotic medications assigned 4 points). The BPI-SF is a self-administered questionnaire developed to assess the severity of pain on a 0-10 categorical scale where 0=no pain, 10=pain as bad as you can imagine. Higher scores indicated worst outcomes. Percentage of Participants Achieving Pain Response assessed using BPI-SF Pain Intensity Score were reported.
Time Frame: Baseline until pain progression, first further anticancer therapy, or data cut-off whichever comes first (maximum duration: up to 141 weeks)
Population: Analysis was performed on subset of ITT population (any participant who had been allocated to a randomized treatment, analyzed according to group allocated) with baseline assessment and at least one post-baseline assessment before any further anti-cancer therapy for specified outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cabazitaxel | Abiraterone Acetate or Enzalutamide
Number analyzed (Participants) | 111 | 109
percentage of participants | 45.9 [36.7 to 55.2] | 19.3 [11.9 to 26.7]

9. Secondary Outcome: Time to Pain Progression
Description: Time to pain progression was defined as the time duration (in months) between the date of randomization and the date of first documented pain progression. Pain progression, in participants with no pain or stable pain at Baseline was defined as increase of >=30% from baseline in the BPI-SF pain intensity score observed at 2 consecutive evaluations >=3 weeks apart without decrease in analgesic usage score or increase in analgesic usage score (calculated from analgesic use data, with non-narcotic medications assigned value of 1 point and narcotic medications assigned 4 points) >=30%. The BPI-SF is a self-administered questionnaire developed to assess the severity of pain on a 0-10 categorical scale where 0=no pain, 10=pain as bad as you can imagine. Higher scores indicated worst outcomes. Analysis was performed by Kaplan-Meier method.
Time Frame: Baseline until pain progression or data cut-off whichever comes first (maximum duration: up to 141 weeks)
Population: Analysis was performed on subset of ITT population (any participant who had been allocated to a randomized treatment, analyzed according to group allocated) with baseline assessment and at least one post-baseline assessment before any further anti-cancer therapy for BPI-SF pain intensity score.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabazitaxel | Abiraterone Acetate or Enzalutamide
Number analyzed (Participants) | 111 | 109
months | NA [NA to NA] — Median, lower and upper limit of CI was not estimable because the curve's upper CI bound had not crossed 50% survival threshold. | 8.5 [4.9 to NA] — Upper limit of CI was not estimable because the curve's upper bound CI had not crossed 50% survival threshold.

10. Secondary Outcome: Number of Symptomatic Skeletal Events (SSE)
Description: SSE was defined as occurrence of a new symptomatic pathological fracture, use of external beam radiation to relieve bone pain, occurrence of spinal cord compression or tumor- related orthopedic surgical intervention.
Time Frame: Baseline until occurrence of first SSE or data cut-off, whichever comes first (maximum duration: up to 141 weeks)
Population: Analysis was performed on ITT population.
Measure: Number; unit: events
Arm/Group | Cabazitaxel | Abiraterone Acetate or Enzalutamide
Number analyzed (Participants) | 129 | 126
events | 24 | 35

11. Secondary Outcome: Time to Symptomatic Skeletal Event
Description: Time to SSE was defined as the time duration (in months) between the date of randomization and the date of occurrence of the first SSE. Analysis was performed by Kaplan-Meier method.
Time Frame: From date of randomization until first SSE, or data cut-off whichever comes first (maximum duration: up to 141 weeks)
Population: Analysis was performed on ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabazitaxel | Abiraterone Acetate or Enzalutamide
Number analyzed (Participants) | 129 | 126
months | NA [20.0 to NA] — Median and upper limit of CI was not estimable because of low number of participants with events. | 16.7 [10.8 to NA] — Upper limit of CI was not estimable because of low number of participants with events.

12. Secondary Outcome: Health-Related Quality of Life (HRQOL): Change From Baseline in Functional Assessment of Cancer Therapy-Prostate (FACT-P) Total Score at Cycle 2, 3, 4, 5, 6, 7, 8 and End of Treatment
Description: Health-related quality of life (HRQOL) evaluation was performed using the FACT-P questionnaire (Version 4). FACT-P was a 39-item participant rated questionnaire that measures the concerns of participants with prostate cancer. It consisted of 5 sub-scales assessing physical well-being (7 items), social/family well-being (7 items), emotional well-being (6 items), functional well-being (7 items), and prostate-specific concerns (12 items). FACT-P total score was the sum of all 5 subscale scores. It ranged from 0 to156 with higher score indicated better quality of life with fewer symptoms. Baseline corresponded to last evaluable assessment before treatment administration.
Time Frame: Baseline, Day 1 of each Cycle 2, Cycle 3, Cycle 4, Cycle 5, Cycle 6, Cycle 7, Cycle 8 and at End of Treatment (any time up to 141 weeks)
Population: Analysis was performed on HRQOL population which included participants who received at least one dose of the study drug and with an evaluable FACT-P questionnaire at baseline and at least one post-baseline evaluable FACT-P. Here 'Number analyzed' signifies participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cabazitaxel | Abiraterone Acetate or Enzalutamide
Number analyzed (Participants) | 108 | 114
score on a scale
  Cycle 2: number analyzed (Participants) | 104 | 106
  Cycle 2 | 2.6 (12.3) | -0.0 (12.4)
  Cycle 3: number analyzed (Participants) | 99 | 94
  Cycle 3 | 2.7 (16.1) | -1.0 (16.8)
  Cycle 4: number analyzed (Participants) | 93 | 77
  Cycle 4 | 2.8 (14.8) | -0.7 (16.8)
  Cycle 5: number analyzed (Participants) | 79 | 56
  Cycle 5 | 2.1 (17.9) | -1.0 (16.1)
  Cycle 6: number analyzed (Participants) | 64 | 39
  Cycle 6 | -3.7 (18.0) | 0.4 (18.6)
  Cycle 7: number analyzed (Participants) | 58 | 33
  Cycle 7 | -2.2 (19.3) | 2.7 (19.9)
  Cycle 8: number analyzed (Participants) | 47 | 25
  Cycle 8 | -4.8 (20.4) | 0.8 (23.0)
  End of treatment: number analyzed (Participants) | 51 | 31
  End of treatment | -6.3 (16.1) | -7.5 (15.7)

13. Secondary Outcome: Change From Baseline in European Quality of Life Working Group Health Status Measure 5 Dimensions, 5 Levels (EQ-5D-5L) Utility Single Index and Visual Analogue Scale (VAS) Scores at Cycle 2, 3, 4, 5, 6, 7, 8 and End of Treatment
Description: EQ-5D was a standardized HRQOL questionnaire consisting of EQ-5D descriptive system and Visual Analogue Scale (VAS). EQ-5D descriptive system comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression measured on 3 levels (no problem, some problems & severe problems) within a particular EQ-5D dimension. 5 dimensional 3-level system was converted into single index utility score. Possible values for single index utility score ranged from -0.594 (severe problems in all dimensions) to 1.0 (no problem in all dimensions) on scale where 1 represented best possible health state. EQ-5D VAS was used to record a participant's rating for his/her current health-related quality of life state and captured on a vertical VAS scale ranging from 0-100, where 0=worst imaginable health state and 100=best imaginable health state, where higher states indicated better outcomes. Baseline corresponded to last evaluable assessment before treatment administration.
Time Frame: Baseline, Day 1 of each Cycle 2, Cycle 3, Cycle 4, Cycle 5, Cycle 6, Cycle 7, Cycle 8 and at End of Treatment (any time up to: 141 weeks)
Population: Analysis was performed on Health status population which included participants who received at least one dose of the study drug and with an evaluable EQ-5D-5L at baseline and with at least one post-baseline evaluable EQ-5D-5L. Here 'Number analyzed' signifies participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cabazitaxel | Abiraterone Acetate or Enzalutamide
Number analyzed (Participants) | 115 | 115
score on a scale
  Cycle 2: VAS: number analyzed (Participants) | 108 | 109
  Cycle 2: VAS | 3.6 (14.4) | 0.9 (14.6)
  Cycle 3: VAS: number analyzed (Participants) | 104 | 94
  Cycle 3: VAS | 4.5 (15.0) | 1.5 (13.4)
  Cycle 4: VAS: number analyzed (Participants) | 100 | 77
  Cycle 4: VAS | 4.6 (16.5) | -1.1 (18.2)
  Cycle 5: VAS: number analyzed (Participants) | 84 | 57
  Cycle 5: VAS | 0.6 (17.1) | 3.2 (17.0)
  Cycle 6: VAS: number analyzed (Participants) | 68 | 39
  Cycle 6: VAS | -1.3 (22.8) | -1.5 (23.1)
  Cycle 7: VAS: number analyzed (Participants) | 60 | 32
  Cycle 7: VAS | 2.9 (18.1) | -0.2 (20.1)
  Cycle 8: VAS: number analyzed (Participants) | 49 | 23
  Cycle 8: VAS | 2.8 (18.0) | 1.2 (19.6)
  End of treatment: VAS: number analyzed (Participants) | 56 | 33
  End of treatment: VAS | -3.3 (19.3) | -5.9 (23.1)
  Cycle 2: Utility Index Score: number analyzed (Participants) | 108 | 109
  Cycle 2: Utility Index Score | 0.026 (0.179) | -0.010 (0.178)
  Cycle 3: Utility Index Score: number analyzed (Participants) | 103 | 94
  Cycle 3: Utility Index Score | 0.041 (0.183) | -0.011 (0.182)
  Cycle 4: Utility Index Score: number analyzed (Participants) | 99 | 79
  Cycle 4: Utility Index Score | 0.051 (0.176) | -0.002 (0.188)
  Cycle 5: Utility Index Score: number analyzed (Participants) | 79 | 59
  Cycle 5: Utility Index Score | 0.027 (0.209) | -0.035 (0.185)
  Cycle 6: Utility Index Score: number analyzed (Participants) | 67 | 42
  Cycle 6: Utility Index Score | 0.015 (0.191) | -0.000 (0.176)
  Cycle 7: Utility Index Score: number analyzed (Participants) | 60 | 34
  Cycle 7: Utility Index Score | 0.029 (0.182) | 0.024 (0.153)
  Cycle 8: Utility Index Score: number analyzed (Participants) | 47 | 24
  Cycle 8: Utility Index Score | 0.008 (0.213) | -0.014 (0.138)
  End of treatment: Utility Index Score: number analyzed (Participants) | 56 | 35
  End of treatment: Utility Index Score | -0.048 (0.188) | -0.079 (0.200)

14. Secondary Outcome: Radiographic Progression-Free Survival (rPFS) in Participants With Presence and Absence of Biomarker
Description: Circulating tumor cell (CTC) counts were considered as biomarker in a liquid biopsy. rPFS in participants with presence and absence of subtypes of CTC biomarker i.e. chromosomal instability (CIN) and neuroendocrine (NE) was reported in this outcome measure. rPFS was defined as: time (in months) from randomization to the first occurrence of any one of following: radiological tumor progressions (RECIST1.1), progression of bone lesions (PCWG2 criteria) or death due to any cause. Progression (RECIST1.1): at least a 20% increase in sum of diameters of target lesions, unequivocal progression of existing non-target lesions. Progression of bone lesions (PCWG2 criteria): first bone scan with >= 2 new lesions compared to Baseline observed <12 weeks from randomization and confirmed by a second bone scan performed >=6 weeks later; first bone scan with >=2 new lesions compared to Baseline observed >=12 weeks from randomization and new lesions were verified on next bone scan >= 6 weeks later.
Time Frame: as for outcome 1
Population: Analysis was performed on subset of participants analyzed according to the treatment group allocated by randomization with evaluable samples.
Measure: Median (Full Range); unit: months
Arm/Group | Cabazitaxel | Abiraterone Acetate or Enzalutamide
Number analyzed (Participants) | 109 | 106
months
  Presence of CIN: number analyzed (Participants) | 27 | 27
  Presence of CIN | 4.2 [2.1 to 11.2] | 4.2 [0.03 to 21.0]
  Absence of CIN: number analyzed (Participants) | 82 | 79
  Absence of CIN | 8.5 [0.03 to 33.1] | 3.4 [0.03 to 28.0]
  Presence of NE: number analyzed (Participants) | 7 | 14
  Presence of NE | 3.0 [2.6 to 11.2] | 3.9 [0.03 to 21.0]
  Absence of NE: number analyzed (Participants) | 102 | 92
  Absence of NE | 8.2 [0.03 to 33.1] | 3.5 [0.03 to 28.0]

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data was collected from Baseline up to 30 days after the last treatment administration (up to 197 weeks), deaths were collected from baseline up to end of study (up to 197 weeks).
Description: Reported AEs were TEAEs i.e., AEs that developed/worsened during the 'on-treatment period' (time from first dose of study drug until 30 days after last administration of study drug) assessed for safety population (i.e., all participants who received at least one dose of study drugs and analyzed according to treatment they actually received). All-Cause Mortality data collected during the study was assessed for all randomized participants. Disease progression related death were not reported as AE.
Groups:
- Enzalutamide or Abiraterone: Participants received either abiraterone acetate 1000 mg orally once daily from Day 1 to Day 21 of each 3 week treatment cycle in combination with prednisone 5 mg orally twice daily; or enzalutamide 160 mg orally once daily continuously from Day 1 to Day 21 of each 3 week treatment cycle, until radiographic disease progression, unacceptable toxicity, or participant's refusal of further study treatment (median duration = 12.5 weeks).
Arm/Group | Cabazitaxel | Enzalutamide or Abiraterone
All-Cause Mortality (participants affected / at risk) | 96/129 | 103/126
Serious Adverse Events (participants affected / at risk) | 49/126 | 50/124
Other Adverse Events (participants affected / at risk) | 114/126 | 104/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabazitaxel (N=126) | Enzalutamide or Abiraterone (N=124)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Hyperfibrinolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Atrial Flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular Block Complete (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac Failure (Cardiac disorders) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea Haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus Paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Asthenia (General disorders) | 3 (4) | 1 (1)
Disease Progression (General disorders) | 4 (4) | 8 (8)
General Physical Health Deterioration (General disorders) | 1 (1) | 2 (2)
Inflammation (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Device Related Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic Infection (Infections and infestations) | 1 (1) | 0 (0)
Perineal Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (5) | 1 (2)
Pulmonary Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Septic Shock (Infections and infestations) | 1 (1) | 0 (0)
Tooth Infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 3 (3)
Urinary Tract Infection Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 0 (0)
Gamma-Glutamyltransferase Increased (Investigations) | 1 (1) | 0 (0)
Platelet Count Decreased (Investigations) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 2 (2)
Neuroendocrine Carcinoma Of The Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oncologic Complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid Artery Stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral Haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive Disorder (Nervous system disorders) | 1 (1) | 0 (0)
Loss Of Consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Paraparesis (Nervous system disorders) | 0 (0) | 1 (1)
Spinal Cord Compression (Nervous system disorders) | 4 (4) | 3 (3)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1) | 0 (0)
Device Dislocation (Product Issues) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 3 (4) | 4 (4)
Haematuria (Renal and urinary disorders) | 1 (1) | 3 (3)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 1 (2)
Pyelocaliectasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 0 (0) | 3 (3)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary Tract Obstruction (Renal and urinary disorders) | 0 (0) | 2 (2)
Pelvic Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive Crisis (Vascular disorders) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabazitaxel (N=126) | Enzalutamide or Abiraterone (N=124)
Anaemia (Blood and lymphatic system disorders) | 38 (75) | 14 (24)
Leukopenia (Blood and lymphatic system disorders) | 8 (12) | 1 (3)
Neutropenia (Blood and lymphatic system disorders) | 28 (35) | 1 (3)
Abdominal Pain (Gastrointestinal disorders) | 10 (12) | 3 (3)
Constipation (Gastrointestinal disorders) | 19 (27) | 13 (18)
Diarrhoea (Gastrointestinal disorders) | 50 (88) | 8 (8)
Nausea (Gastrointestinal disorders) | 29 (49) | 26 (31)
Stomatitis (Gastrointestinal disorders) | 10 (13) | 2 (3)
Vomiting (Gastrointestinal disorders) | 16 (21) | 14 (18)
Asthenia (General disorders) | 33 (69) | 26 (37)
Fatigue (General disorders) | 36 (65) | 21 (27)
Oedema Peripheral (General disorders) | 10 (13) | 11 (12)
Pain (General disorders) | 8 (8) | 6 (7)
Pyrexia (General disorders) | 7 (10) | 7 (7)
Urinary Tract Infection (Infections and infestations) | 10 (10) | 4 (4)
Weight Decreased (Investigations) | 5 (6) | 7 (7)
Decreased Appetite (Metabolism and nutrition disorders) | 16 (21) | 19 (21)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (8) | 7 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (14) | 20 (35)
Back Pain (Musculoskeletal and connective tissue disorders) | 20 (22) | 27 (41)
Bone Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 7 (7)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 6 (7) | 13 (18)
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (15) | 9 (10)
Dysgeusia (Nervous system disorders) | 15 (18) | 5 (7)
Neuropathy Peripheral (Nervous system disorders) | 8 (11) | 3 (3)
Polyneuropathy (Nervous system disorders) | 8 (12) | 0 (0)
Haematuria (Renal and urinary disorders) | 18 (27) | 5 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 3 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (7) | 0 (0)
Hypertension (Vascular disorders) | 5 (12) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT02485691/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT02485691/SAP_001.pdf